CLINICAL TRIAL: NCT03638804
Title: 89Zr-labeled KN035 PET Imaging in Patients With PD-L1positive Advanced Solid Tumors
Brief Title: 89Zr-KN035 PET Imaging in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: MITRO Biotech Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Miao Liyan, Professor, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMS-2017-007-a
Record Dates: First submitted 2018-07-23; First posted 2018-08-20 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Solid Tumor, Adult
Keywords: 89Zr; PD-L1; KN035; PET

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 89Zr-KN035 injection (Experimental)
  Interventions: Diagnostic Test: 89Zr-KN035

INTERVENTIONS:
Diagnostic Test: 89Zr-KN035 — Single injection of 89Zr labeled KN035 in subjects to observe KN035 affinity in PD-L1 expressed Solid tumors by using PET imaging.

SUMMARY:
This is a single arm study by using 89Zr-labeled KN035 (89Zr-KN035) PET imaging to evaluate the biodistribution and target lesion uptake of 89Zr-KN035 in patients with PD-L1 positive advanced solid tumors.

DETAILED DESCRIPTION:
The overall purpose of the study is to evaluate the biodistribution and target lesion uptake of 89Zr-KN035 in patients with PD-L1 positive advanced solid tumors by using PET imaging. Safety will be observed after 89Zr-KN035 injection, and radiation dosimetry of 89Zr-KN035 will be calculated.

ELIGIBILITY:
Inclusion Criteria (main):

1. Patients voluntarily signed informed consent;
2. Age 18-75, male or female;
3. Patients diagnosed with locally advanced or metastatic solid tumors by histopathology or cytology;
4. Patients with biopsy-proven PD-L1 positive;
5. ECOG score ≤ 0~1; Life expectancy of at least 3 months;
6. Women of childbearing age are required to receive serum pregnancy tests, and only those who have a negative pregnancy test for eligible subjects.

Exclusion Criteria(main):

1. Currently or within the first 28 days before the first dose to participate in another therapeutic clinical trial. If participating in a non-interventional clinical trial, it is not be excluded.
2. Patients with systemic or locally severe infections (CTCAE ≥ 2);
3. Patients with allergies or allergies to any component of the imaging agent or antibody;
4. Patients who cannot undergo PET/CT imaging;
5. Intolerance of intravenous administration, as well as difficulties in venous blood collection (If having the medical history of fainting during acupuncture, and blood phobia);
6. Symptomatic congestive heart failure (NYHA class II-IV) or symptomatic or poorly controlled arrhythmia;
7. Patients have significant QT/QTC interval prolongation during the screening period;
8. Received anti-tumor therapy (including but not limited to chemotherapy, radiotherapy, biological therapy) within 4 weeks prior to first dose;
9. Patents have not recovered to CTCAE grade 0 or 1 from the adverse events due to cancer therapeutics administered;
10. Previously received CD137 agonist or immune checkpoint blocking therapy;
11. Patients with diabetes who have a fasting blood glucose greater than 10 mmol/L;
12. HIV antibody positive, active hepatitis B/C, and TB positive;
13. Patients are regular users (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol);
14. Patients with symptomatic ascites, pleural effusion, or hydropericardium;
15. Pregnant or lactating women, or planning to become pregnant or have children during this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Description of regions of interest (ROI) 89Zr-KN035 by measuring standardized uptake value (SUV) on 89Zr-KN035 PET scans | 6 months

SECONDARY OUTCOMES:
Number of adverse events as assessed by CTCAE v4.03 | 6 months
  All adverse events will be assessed by CTCAE v 4.03 and evaluated if treatment-related or not.
Number of changes in laboratory test results as accessed by CTCAE v4.03 | 6 months
  Laboratory tests (blood, urine) will be conducted by time. Significant changes will be assessed by CTCAE v 4.03.
Number of changes in vital signs as accessed by CTCAE v4.03 | 6 months
  Vital signs (heart rate, respiratory rate, blood pressures and body temperature) data will be collected by time. Significant changes will be assessed by CTCAE v4.03.

OTHER OUTCOMES:
Maximum serum concentration of 89Zr-KN035 (Cmax) | 6 months
  Blood samples will be collected and assessed by timepoints.
Time to Maximum Concentration of 89Zr-KN035 (Tmax) | 6 months
  Blood samples will be collected and assessed by timepoints.
Calculation of radiation dosimetry of 89Zr-KN035 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Liyan Miao, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University; Jianan Huang, PhD, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China